CLINICAL TRIAL: NCT01299532
Title: An Open, Multi-center Study Evaluating Efficacy and Safety of Macrolane VRF30 for Enhancement of the Shape and Fullness of the Female Breast
Brief Title: Macrolane VRF30 for Enhancement of Shape and Fullness of Female Breast
Acronym: COBRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 31GB0801
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2011-02

CONDITIONS: Breast Enhancement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Macrolane VRF30 (Experimental)
  Interventions: Device: Macrolane VRF30

INTERVENTIONS:
Device: Macrolane VRF30 — Device: Macrolane VRF30 (stabilized hyaluronic acid of non-animal origin) Treatment: Initial injection of a maximum of 120 ml/breast. Re-injection of a maximum of 120 ml/breast in a subgroup of subjects.

SUMMARY:
This is an open, multi-center, non comparative study to evaluate the safety and efficacy of Macrolane VRF30 in the female breast. 71 subjects have received initial treatment with a maximum of 120 ml of Macrolane VRF30 per breast. 22 patients have received a re-injection (max 120 ml/breast) of Macrolane nine months after initial treatment. Patients are followed for 24 months after last treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 25 and 60 years with small breasts seeking enhancement of the shape and fullness of the breast

Exclusion Criteria:

* Unreasonable expectations as regards the increase in breast volume
* Any medical conditions that may interfere in any way.

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2008-11; Primary Completion 2010-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Perceived improvement of shape and fullness of the female breast compared to baseline as judged by the subject using GEIS. | 6 months

SECONDARY OUTCOMES:
To evaluate the safety as documented by physical examination, mammography, ultrasonography and by adverse events reported. | 24 months
To evaluate adverse experiences occurring during the first 2 weeks post treatment as recorded in the diary. | 2 weeks
to study the implant duration and localization as documented by MRI. | 24 months
to evaluate esthetic improvement of shape and fullness as judged by an independent evaluator, by the investigator and by the subject using GEIS. | 24 months
to evaluate the subjects satisfaction with her breast and general appearance using a subject questionnaire. | 24 months
to evaluate pain experience during injection under local anesthesia. | during injection
To evaluate any difficulties with the interpretation of the mammography image(s)or ultrasonography due to the presence of the implant 24 months after the initial treatment | 24 months
Re-treatment phase: To evaluate the safety documented by physical examination and by adverse events reported up to 24 months after re-treatment and by mammography and ultrasonography examinations 15 and 39 months after re-treatment. | 39 months
Re-treatment phase: To evaluate any difficulties with the interpretation of the mammography image(s) or ultrasonography due to the presence of the implant 24 and 48 months after the initial treatment (15 and 39 months after the re-treatment). | 48 months
Re-treatment phase: To evaluate adverse experiences occurring during the first 2 weeks post re-treatment as recorded in the diary. | 2 weeks
Re-treatment phase: To study the implant duration and localization as documented by MRI up to 24 months after re-treatment. | 24 months
Re-treatment phase: To evaluate esthetic improvement of shape and fullness as judged by an independent evaluator, by the investigator and by the subject using GEIS up to 24 months after re-treatment. | 24 months
Re-treatment phase: To evaluate, up to 24 months after re-treatment, the subjects satisfaction with her breast and general appearance using a subject questionnaire. | 24 months
Re-treatment phase: To evaluate pain experience during re-injection under local anaesthesia. | During re-injection
Re-treatment phase: To evaluate if there are differences in esthetic improvement, subject satisfaction and implant duration, after re-treatment compared to after initial treatment. The visits up to 9 months will be compared. | 9 months
Re-treatment phase: To compare esthetic improvement, subject satisfaction and implant duration at 24 months after last treatment between subjects that have received only one treatment and subjects that have received re-treatment. | 24 months
Re-treatment phase: To compare esthetic improvement, subject satisfaction and implant duration at 12 and 24 months after initial treatment between subjects that have received only one treatment and subjects that have received re-treatment. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Per Hedén, M.D., Ph.D., Principal Investigator — Akademikliniken, Stockholm, Sweden
Locations (5):
- France (2):
  - Sainte Anne, Paris
  - L'Institute du Sein, Paris
- Sweden (3):
  - Plastikkirurggruppen, Stockholm
  - Akademikliniken, Stockholm
  - Proforma Clinic, Stockholm